CLINICAL TRIAL: NCT06570343
Title: Analgesic Efficacy of Intrathecal Fentanyl-Morphine Combination Versus Morphine Alone for Intraoperative Pain During Elective Cesarean Delivery: a Randomized Clinical Trial
Brief Title: Analgesic Efficacy of Intrathecal Fentanyl-Morphine Combination Versus Morphine Alone for Intraoperative Pain During Elective Cesarean Delivery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2407-091-1553
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Intraoperative Pain
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl-Morphine (Experimental): Spinal anesthesia with heavy bupivacaine, fentanyl and morphine
  Interventions: Drug: Fentanyl-Morphine
- Morphine (Active Comparator): Spinal anesthesia with heavy bupivacaine and morphine
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Fentanyl-Morphine — Intrathecal injection of bupivacaine, fentanyl and morphine
  Arms: Fentanyl-Morphine
Drug: Morphine — Intrathecal injection of bupivacaine and morphine
  Arms: Morphine

SUMMARY:
Pregnant women scheduled for elective cesarean sections under spinal anesthesia are randomly assigned to two groups: 1) the Fentanyl-Morphine (FM) group, and 2) the Morphine (M) group. In addition to 11.5 mg of bupivacaine, the FM group receives 15 μg of fentanyl and 50 μg of morphine intrathecally, while the M group receives 50 μg of morphine intrathecally. The incidence of intraoperative pain with a Numerical Rating Scale (NRS) score of 4 or higher is compared between the two groups to evaluate the analgesic effects of combined intrathecal fentanyl-morphine therapy versus morphine alone.

ELIGIBILITY:
Inclusion Criteria:

* Parturients of gestational age > 37 weeks, scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Contraindication to spinal anesthesia
* Any sign of onset of labor
* Emergency cesarean section
* Body weight < 40 kg or > 120 kg
* Height < 140 cm or > 190 cm
* Severe underlying cardiovascular disease
* Known fetal anomaly
* Preeclampsia
* History of hypersensitivity to fentanyl or morphine
* Chronic opioid use

Ages: 19 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative pain | From first skin incision to end of surgery
  Incidence of intraoperative pain of NRS (numeric rating scale) score of 4 or higher

SECONDARY OUTCOMES:
Time of occurence of intraoperative pain | From first skin incision to end of surgery
  Time of occurence of intraoperative pain of NRS (numeric rating scale) score of 4 or higher
Incidence of intraoperative rescue analgesic administration | From first skin incision to end of surgery
  Incidence of intraoperative rescue analgesic administration
Total amount of intraoperative opioid rescue analgesic administration | From first skin incision to end of surgery
  Total amount of intraoperative opioid rescue analgesic administration (morphine mg equivalent)
Total amount of intraoperative non-opioid rescue analgesic administration | From first skin incision to end of surgery
  Total amount of intraoperative non-opioid rescue analgesic administration (mg)
Intraoperative pain characteristics | From first skin incision to end of surgery
  Intraoperative pain characteristics
Conversion to general anesthesia | From first skin incision to end of surgery
  Conversion to general anesthesia
Preoperative anxiety | On the day before surgery
  Preoperative anxiety (APAIS, Amsterdam Preoperative Anxiety and Information Score)
Preoperative anxiety | On the day of surgery
  Preoperative anxiety (APAIS, Amsterdam Preoperative Anxiety and Information Score)
Total amount of postoperative opioid analgesic administered | From end of surgery to 24 hours after end of surgery
  Total amount of postoperative opioid analgesic administered (morphine mg equivalent)
Incidence of intraoperative nausea/vomiting | From induction to end of surgery
  Incidence of intraoperative nausea/vomiting
Incidence of postoperative nausea/vomiting | From end of surgery to 24h post-surgery
  Incidence of postoperative nausea/vomiting
Incidence of intraoperative shivering | From induction to end of surgery
  Incidence of intraoperative shivering
Incidence of intraoperative hypotension | From induction to end of surgery
  Incidence of intraoperative hypotension (MBP<65 mmHg)
Incidence of intraoperative pruritus | From induction to end of surgery
  Incidence of intraoperative pruritus
Incidence of postoperative pruritus | From end of surgery to 24h post-surgery
  Incidence of postoperative pruritus
Immediate post-operative patient satisfaction | At the end of surgery
  Immediate post-operative patient satisfaction on intraoperative analgesia
Obstetric Quality of Recovery-11K score | At 24 hours post-surgery
  Obstetric Quality of Recovery-11K score
Time of first postoperative pain | From end of surgery to 24 hours post-surgery
  Time of first postoperative pain
Pain score at 8 hours post-surgery | at 8 hours post-surgery
  Pain score at 8 hours post-surgery (NRS, numeric rating scale pain score, 0: no pain; 10: worst imaginable pain)
Pain score at 16 hours post-surgery | at 16 hours post-surgery
  Pain score at 16 hours post-surgery (NRS, numeric rating scale pain score, 0: no pain; 10: worst imaginable pain)
Pain score at 24 hours post-surgery | at 24 hours post-surgery
  Pain score at 24 hours post-surgery (NRS, numeric rating scale pain score, 0: no pain; 10: worst imaginable pain)
Pain score at 2 hours post-surgery | at 2 hours post-surgery
  Pain score at 2 hours post-surgery (NRS, numeric rating scale pain score, 0: no pain; 10: worst imaginable pain)
Incidence of postoperative hypotension | From end of surgery to 24 hours post-surgery
  Incidence of postoperative hypotension (MBP<65 mmHg)
Incidence of postoperative shivering | From end of surgery to 24 hours post-surgery
  Incidence of postoperative shivering
24-hour post-operative patient satisfaction | at 24 hours post-surgery
  24-hour post-operative patient satisfaction on postoperative analgesia

IPD SHARING:
Plan to Share IPD: No